CLINICAL TRIAL: NCT06627088
Title: A Phase 1, Open-label, Two-part Study of the Absorption, Metabolism, Excretion, and Bioavailability of LY4100511 (DC-853) Following Administration of [14C]-LY4100511 in Healthy Male Participants
Brief Title: A Study of LY4100511 (DC-853) Mass Balance and Absolute Bioavailability of LY4100511 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27109; J5C-MC-FOAE (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2024-09-12; First posted 2024-10-04 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: LY4100511; DC-853

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A LY4100511 (tablet formulation) and [14C]-LY4100511 capsule (Experimental): Participants will receive a single oral dose 1 or dose 2 unlabeled LY4100511 (tablet formulation) administered with a dose 1 [14C]-LY4100511 capsule containing approximately 100 µCi (3.7 MBq) of radioactivity in the fasted state
  Interventions: Drug: LY4100511 (DC-853); Drug: [14C]-LY4100511 (DC-853) Administered oral dose
- Part B LY4100511 (tablet formulation) and [14C]-LY4100511 (Experimental): Participants will receive a single oral dose 1 or dose 2 unlabeled LY4100511 (tablet formulation) in the fasted state, followed by a single intravenous (IV) dose of of [14C]-LY4100511, containing ≤1 μCi (≤37 kBq) of radioactivity, administered as an infusion.
  Interventions: Drug: LY4100511 (DC-853); Drug: [14C]-LY4100511 (DC-853)

INTERVENTIONS:
Drug: LY4100511 (DC-853) — Administered oral dose
  Arms: Part A LY4100511 (tablet formulation) and [14C]-LY4100511 capsule
Drug: [14C]-LY4100511 (DC-853) Administered oral dose — Administered oral dose
  Arms: Part A LY4100511 (tablet formulation) and [14C]-LY4100511 capsule
Drug: LY4100511 (DC-853) — Administered oral dose
  Arms: Part B LY4100511 (tablet formulation) and [14C]-LY4100511
Drug: [14C]-LY4100511 (DC-853) — Administered IV infusion
  Arms: Part B LY4100511 (tablet formulation) and [14C]-LY4100511

SUMMARY:
The study has two parts, Part A and Part B. The purpose of Part A is to determine the absorption, metabolism, and excretion (AME) of [14C]-LY4100511 and to characterize and determine the metabolites present in plasma, urine, and feces in healthy male participants after a single oral dose of LY4100511. The purpose of Part B is to determine the absolute bioavailability of LY4100511 in humans, to further analyze the rate and routes of excretion, including the mass balance, and to further investigate the pharmacokinetics (PK) of [14C]-LY4100511, LY4100511, and TRA.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kilogram per square meter (kg/m2), inclusive, and a body weight of ≥50 kilogram (kg)
* In good health and determined by no clinically significant finding from medical history, 12-lead ECG and vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia, e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin is not acceptable) at screening and check-in, and from the physical examination at check-in, as assessed by the Investigator or designee
* History of a minimum of 1 bowel movement per day.
* Able to provide a fecal sample between check-in on Day-2 and oral dosing on Day 1.

Exclusion Criteria:

* Have a 12-lead ECG abnormality that, in the opinion of the Investigator

  * increases the risks associated with participating in the study
  * may confound ECG data analysis
  * a QTcF & > 450 msec
  * short PR interval & <120 msec or PR interval >220 msec
  * second- or third-degree atrioventricular block
  * intraventricular conduction delay with QRS 120 msec
  * right bundle branch block
  * left bundle branch block, or
  * Wolff Parkinson-White syndrome.
* Have a current or recent acute, active infection (for example, for at least 30 days before screening and up to check-in, participants must have no symptoms or signs of infection in the absence of any anti-infective treatment).
* Had any malignancy within the past 5 years. Exceptions: successfully treated basal cell skin carcinoma or squamous cell skin carcinoma, with no evidence of recurrence or metastatic disease within the 3 years prior to baseline.
* Are immunocompromised.
* Have inflammatory bowel disease (IBD)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — individuals assigned male at birth
Enrollment: 24 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Part A: Total Radioactivity Recovery and Excretion (TRA) | Up until Day 15
  Total radioactivity recovery and excretion (fet1-t2 and Aet1-t2) in urine and feces (and vomitus, if available)
Part A: Pharmacokinetic (PK): Area Under the Concentration from Time 0 to Infinity (AUC0-∞) for [14C] LY4100511 | Up until Day 15
Part A: Pharmacokinetic (PK): Area Under the Concentration from Time 0 to Infinity (AUC0-∞) for LY4100511 | Up until Day 15
Part A: Pharmacokinetic (PK): Area Under the Concentration from Time 0 to Infinity (AUC0-∞) for TRA | Up until Day 15
Part A: PK Area Under Concentration from 0 to Last Measurable Concentration (AUC0-tlast) for [14C] LY4100511 | Up until Day 15
Part A: PK Area Under Concentration from 0 to Last Measurable Concentration (AUC0-tlast) for LY4100511 | Up until Day 15
Part A: PK Area Under Concentration from 0 to Last Measurable Concentration (AUC0-tlast) for TRA | Up until Day 15
Part A: PK Maximum Observed Plasma Concentration (Cmax) for [14C] LY4100511 | Up until Day 15
Part A: PK Maximum Observed Plasma Concentration (Cmax) for LY4100511 | Up until Day 15
Part A: PK Maximum Observed Plasma Concentration (Cmax) for TRA | Up until Day 15
Part A: PK Time to Maximum Observed Plasma Concentration (tmax) for [14C] LY4100511 | Up until Day 15
Part A: PK Time to Maximum Observed Plasma Concentration (tmax) for LY4100511 | Up until Day 15
Part A: PK Time to Maximum Observed Plasma Concentration (tmax) for TRA | Up until Day 15
Part A: PK Terminal Elimination Half Life (t1/2) for [14C] LY4100511 | Up until Day 15
Part A: PK Terminal Elimination Half Life (t1/2) for LY4100511 | Up until Day 15
Part A: PK Terminal Elimination Half Life (t1/2) for TRA | Up until Day 15
Part A: Urinary Recovery and Excretion of TRA (Aet1-t2) | Up until Day 15
Part A: Urinary Recovery and Excretion of [14C] LY4100511 (Aet1-t2) | Up until Day 15
Part A: Renal clearance of [14C] LY4100511 (CLR) | Up until Day 15
Part B: Pharmacokinetic (PK): absolute bioavailability (Fabs) of LY4100511 | Up until Day 6
Part B: Recovery of TRA in urine and feces | Up until Day 6
Part B: Recovery of [14C]-LY4100511 in feces (Aet1-t2) following IV dosing | Up until Day 6
Part B: Recovery of [14C]-LY4100511 in urine (Aet1-t2) following IV dosing | Up until Day 6
Part B: PK Area Under Concentration from 0 to Last Measurable Concentration (AUC0-tlast) of LY4100511 following IV dosing | Up until Day 6
Part B: PK Maximum Observed Plasma Concentration (Cmax) of LY4100511following IV dosing | Up until Day 6
Part B: PK Time to Maximum Observed Plasma Concentration (tmax) of LY4100511following IV dosing | Up until Day 6
Part B: PK Terminal Elimination Half Life (t1/2) following IV dosing | Up until Day 6
Part B: PK Clearance (CL) following IV dosing | Up until Day 6
Part B: PK renal clearance (CLr) following IV dosing [Time Frame: Up until Day 6] | Up until Day 6

SECONDARY OUTCOMES:
Number of Participants with One or More Adverse Events (AEs), and Serious Adverse Events (SAEs) considered by the investigator to be related to study drug administration | Up until Day 8
  A summary of AEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events Module.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No